CLINICAL TRIAL: NCT02031328
Title: Two StereoTactic Ablative Adaptive Radiotherapy Treatments for Localized Prostate Cancer
Acronym: 2STAR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Andrew Loblaw, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 312-2013
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prostate Adenocarcinoma
Keywords: prostate; radiation; stereotactic body radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Ablative Radiation (Experimental): Stereotactic Ablative Radiation 26 Gy in 2 fractions, once weekly to prostate
  Interventions: Radiation: Stereotactic Ablative Radiation

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiation

SUMMARY:
You have been asked to consider participating in the study because you have a cancer of the prostate, which is to be treated with external beam radiation. You have chosen or felt not to be a good candidate for just watching your cancer. As your doctor has informed you, this involves delivering small amounts of radiation daily over several weeks. Normally, a small field directed to the prostate gland is given for 7.5 - 8 weeks. In total, 39 days of radiation are delivered. There is now growing evidence that prostate cancer cells may be killed more effectively if higher doses of radiation are delivered everyday (known as hypofractionation). However, the downside to such a strategy is the potential to cause more side effects because normal organs (such as the rectum and bladder) are also exposed to the higher doses. Stereotactic ablative radiotherapy (SABR) is a high-precision technique which has the ability to deliver radiation in a more focused manor, meaning that the radiation dose can be "sculpted" to the prostate gland, while minimizing the amount of radiation to the bladder and rectum.

A certain amount of movement of the prostate normally occurs within the body. To make sure that the prostate will not be missed, a margin of tissue around the prostate also needs to be treated. Although a wide margin will ensure that the prostate is included, it will also cause more normal tissue to receive high doses of radiation. This, in turn, would result in more side effects. To reduce the margin needed around the prostate, and side effects, tiny gold seeds measuring 3.0 x 1.2mm will be inserted into the prostate which can be seen using a special type of X-Ray camera called a portal imager during treatment. This will allow for targeting of the prostate gland more precisely so that a significantly smaller margin of normal tissue will need to be treated. By using gold seeds in conjunction with SABR, there is the potential to safely deliver a more intensive dose of radiation to the prostate gland without increasing the amount of side effects.

In other studies where shorter and more intense courses of radiation have been given using similar high-precision techniques, the side effects of treatment have indeed been no worse than the usual techniques. Over the last 7 years, Sunnybrook researchers have treated over three hundred prostate cancer patients on various research protocols with SABR. In those protocols, patients received 5 SBRT treatments over 29 days and this is currently being compared to 5 SBRT treatments over 11 days in an ongoing randomized study. In the United States, several groups have investigated the 5 SBRT approach in 11 days or less and early findings suggest a good tolerance.

The study is being done to determine the side effects, quality of life and efficacy of 2-fraction adaptive SBRT technique (2STAR) in the treatment of low and intermediate risk prostate cancer. All participants will receive the same dose and fractionation scheme.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Men >18 years
* Histologically confirmed prostate adenocarcinoma (centrally reviewed)
* Low and intermediate risk prostate cancer, defined as clinical stage T1-2b, Gleason Score less than/equal to 7, and PSA less than 20 ng/mL (low risk patients will have refused or felt to be inappropriate for active surveillance)

Exclusion Criteria:

* Androgen deprivation therapy (LHRH-agonists or antiandrogens)>6 mo
* Prior pelvic radiotherapy
* Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* Diagnosis of bleeding diathesis
* Large prostate (>90cm3) on imaging
* Immunosuppressive medications
* Inflammatory bowel disease
* Presence of a hip prosthesis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2014-09-12 (Actual); Study Completion 2024-09-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 5 years
  To determine the prostate-specific quality of life (QOL) using the Expanded Prostate Cancer Index Composite (EPIC) 37 questionnaire for patients undergoing a 2 fraction SBRT protocol. QOL using the Expanded Prostate Cancer Index Composite (EPIC) will be obtained at baseline, weeks 1, 4, 12, month 6 and every 6 months until year 5.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Loblaw, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Science Centre Odette Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ong WL, Cheung P, Chung H, Chu W, Detsky J, Liu S, Morton G, Szumacher E, Tseng CL, Vesprini D, Davidson M, Ravi A, McGuffin M, Zhang L, Mamedov A, Deabreu A, Kulasingham-Poon M, Loblaw A. To Boost or Not to Boost: Pooled Analyses From 2-Fraction SABR Trials for Localized Prostate Cancer. Int J Radiat Oncol Biol Phys. 2023 Dec 1;117(5):1153-1162. doi: 10.1016/j.ijrobp.2023.06.250. Epub 2023 Jul 5. PMID 37419394